CLINICAL TRIAL: NCT03233152
Title: A Phase I/II Clinical Trial on the Per-operative Intratumoral Administration of Myeloid Dendritic Cells Plus Ipilimumab and Nivolumab, Followed by Repeated Intracavitary Plus Intravenous Administration of Nivolumab in Patients With Recurrent Glioblastoma
Acronym: GlitIpNi
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Bart Neyns, Head of Medical Oncology, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-BN-002
Record Dates: First submitted 2017-07-17; First posted 2017-07-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma
Keywords: recurrence
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Ipilimumab; Solutions; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ipilimumab + nivolumab + CD1c (BDCA-1)+ myDC and CD141 (BDCA-3)+ myDC (Experimental): Phase I CD1c(BDCA-1)+/CD141(BDCA-3)+ myDC dose escalation (: 3 predefined dose levels) part of the study: to document the safety of peroperative injection of an escalating number of autologous CD1c(BDCA-1)+/CD141(BDCA-3)+ myDC plus IT injection of nivolumab and ipilimumab, following tumor resection.
  Phase II part of the study: to document the anti-tumor activity of peroperative injection of a defined number of autologous CDC1(BDCA-1)+/CD141(BDCA-3)+myDC. Ipilimumab (YervoyTM, 50 mg/10 mL) and Nivolumab (OpdivoTM, 40 mg/4mL solution) will be administered peroperatively at a dose of injection of 10 mg (2 ml of YervoyTM, 50 mg/10mL vial). as well as intracavitary on days 15, 29, 43, 57, 71, 85, 99, 113, 127, 141, 155 and 169.
  10 mg Nivolumab by the intravenous route will be administered by a 15 minutes intravenous infusion on days 15, 29, 43, 57, 71, 85, 99, 113, 127, 141, 155 and 169. (or up to ± 3 days before or after the scheduled date if necessary).
  Interventions: Drug: Ipilimumab (YervoyTM, 50 mg/10 mL solution); Drug: Nivolumab (OpdivoTM, 40 mg/4mL solution); Biological: Autologous CD1c(BDCA-1)+ /CD141(BDCA-3)+ myDC

INTERVENTIONS:
Drug: Ipilimumab (YervoyTM, 50 mg/10 mL solution) — Ipilimumab will be administered by at the end of the neurosurgical resection procedure at a dose of injection of 10 mg (: 2 ml of YervoyTM, 50 mg/10mL vial).
  Injections will be performed manually using a 100 μ-liter dispensing syringe. Twenty needle tracks will dispense the ipilimumab solution within the brain tissue lining the resection cavity. The region suspect on preoperative MRI of the brain to be invaded by glioblastoma cells but not amenable to safe resection will be targeted by adjacent needle tracks through which up to 2 cm of depth a volume of 100 μl per needle track will be injected (: in total 20 needle tracks will be performed). This methodology has been applied previously within the context of phase III clinical trials with sitimagene ceradenovec.
  Other Names: Nivolumab (OpdivoTM, 40 mg/4 mL solution)
Drug: Nivolumab (OpdivoTM, 40 mg/4mL solution) — First administration of 10 mg of nivolumab by the intravenous route should be administered within 24 hours prior to the planned neurosurgical resection. Administrations of 10 mg nivolumab (OpdivoTM, 40 mg/4mL solution) will be by a 15 minutes intravenous infusion on days 15, 29, 43, 57, and 71 (or up to ± 3 days before or after the scheduled date if necessary).
Biological: Autologous CD1c(BDCA-1)+ /CD141(BDCA-3)+ myDC — Autologous CD1c(BDCA-1)+/CD141(BDCA-3)+ myDC will be isolated from PBMC obtained from the leukapheresis. These are injected in the neighbouring brain tissue post tumor resection.

SUMMARY:
Phase I/II clinical trial on the per-operative intra-tumoral administration of myeloid dendritic cells plus ipilimumab and nivolumab, followed by repeated intracavitary administration of ipilimumab and nivolumab plus intravenous administration of nivolumab in patients with recurrent glioblastoma.

The aim of this clinical trial is to exploit the potential synergy of combined intra-tumoral CTLA-4 and autologous CD1c(BDCA-1)+/CD141(BDCA-3)+ myDC and systemic PD-1 blockade while minimizing the risk for increased immune-related toxicity by intratumoral administration of the CTLA-blocking mAb ipilimumab following the resection of the recurrent glioblastoma.

DETAILED DESCRIPTION:
Nivolumab (OpdivoTM, BMS), a human IgG-4 mAb that blocks the Programmed cell death protein 1 (PD-1, CD279) has demonstrated anti-tumor activity in patients with various solid- and hematological neoplasms. Nivolumab has been registered by EMA and/or FDA for the treatment of patients with advanced melanoma, renal cell carcinoma (RCC), non-small cell lung cancer (NSCLC), and Hodgkin lymphoma. In a phase I dose escalation clinical trial, receptor blockade of PD-1 by nivolumab on circulating lymphocytes was maximal at a dose of 0,3 mg/kg. In patients with advanced melanoma nivolumab had a comparable tumor response rate at a dose range of 0.1 to 10 mg/kg q2wks. Nivolumab was further developed at a dose of 3 mg/kg q2wks and improved the overall survival of patients with advanced melanoma, NSCL, RCC and HNSCC.

Ipilimumab (YervoyTM, BMS), a human IgG-1 anti-CTLA-4 monoclonal antibody improves the overall survival of patients with advanced melanoma; and the relapse-free survival after complete resection of high-risk stage III melanoma. Animal models have established the safety and efficacy of intra-tumoral administration of ipilimumab. An intratumoral dose of CTLA-4 blocking mAb administered at a ratio of [1:100] compared to intravenous dosing was found to result in equivalent anti-tumor effect and was associated with less systemic toxicity.

Combined treatment with ipilimumab (3 mg/kg q3wks x4) plus nivolumab (1 mg/kg q3 wks x4 followed by 3 mg/kg q2 wks) further increases the tumor response rate and progression-free survival of patients with advanced melanoma and has been registered by EMA and FDA; this combination therapy is associated with a higher incidence of immune related adverse events. Nivolumab and ipilimumab have distinct immunological mechanisms that can be revealed by analyzing TCR usage in blood lymphocytes.

Preliminary safety and activity of nivolumab and its combination with ipilimumab in recurrent glioblastoma (CHECKMATE-143) were presented at the 2015 and 2016 ASCO Annual meetings (20 pts were treated, 10 in each arm). [15] All nivolumab related AEs were grade 1 or 2. Eight (80%) nivolumab plus ipilimumab treated patients experienced grade 3/4 AEs. Drug-related AEs leading to discontinuation occurred only in nivolumab plus ipilimumab patients (n = 5; 50%), including colitis, cholecystitis, diabetic ketoacidosis, confusion, and increased lipase. There were no drug-related deaths. Based on these experiences, the sponsor (BMS) decided to further investigate nivolumab as a mono-therapy in patients with recurrent- and newly diagnosed glioblastoma (CA209-143; CA209-498 and CA209-548). Antitumor activity of nivolumab has recently been established in children with recurrent glioblastoma that is characterized by biallelic mismatch repair deficiency.

Recent insight into the interplay of myeloid and lymphoid cells in the tumor microenvironment (TME) has indicated a pivotal role for myeloid dendritic cells (myDC) as key-mediators in mediating an adaptive anti-tumor immune response and also in "re-licensing" antitumoral CTL within the TME. Even when present in very low numbers, these cells play an essential role in "re-licensing" of antitumoral CTL within the TME. (Broz, Binnewies et al. 2014) CD1c (BDCA-1)+ myDC and CD141 (BDCA-3)+ myDC are able to capture tumor antigens in vivo. Through the cross presentation of tumor antigens CD1c (BDCA-1)+ myDC and CD141 (BDCA-3)+ myDC can coordinate an effective antitumoral T-cell response.

ELIGIBILITY:
1. Subjects must have signed and dated an approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care
2. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study.
3. Histopathological diagnosis of glioblastoma (= WHO grade IV glioma of the central nervous system); both patients with "de novo" and "secondary" glioblastoma are eligible; patients who have histological proof of a lower-grade glioma (WHO grade I, II or III) and have evidence for transformation to WHO-grade IV glioma on imaging of the brain (gadolinium enhancement, areas of necrosis) are eligible for study participation;
4. Diagnosis of glioblastoma recurrence and/or progression following prior treatment with surgery consisting of a total or partial tumor resection, radiation therapy and temozolomide chemotherapy (recurrence/progression is defined as significant [according to the investigators assessment] growth and/or recurrence of the glioblastoma tumor mass on sequential MRI of the brain);
5. The following disease characteristics should be present:

   1. Presence of a measurable tumor lesion that is characterized by gadolinium enhancement on T1-MRI of the brain (with a longest diameter of > 10 mm and a perpendicular diameter of >5mm).
   2. No evidence of clinically relevant spontaneous intra-tumor hemorrhage on baseline MRI imaging or in the prior disease history
6. No ventriculo-peritoneal drain
7. No contraindication for evaluation by gadolinium enhanced MRI, FET-PET of the brain or whole-body contrast enhanced CT;
8. ECOG performance status score of 0, 1 or 2;
9. An interval of at least 4 months (: 16 weeks) after the end of postoperative radiation therapy for glioblastoma unless progression is confirmed on an MRI of the brain obtained > 4 week after the first observation of progression; and with an interval of at least 4 weeks after the last administration of temozolomide;
10. Male or female, 18 years of age or older;
11. Resolution of all acute treatment related adverse effects of prior surgical procedures, radiotherapy and temozolomide to NCI CTCAEv4.0 grade 0 or 1 except for alopecia;
12. Adequate organ function as defined by the following criteria:

    1. Total serum bilirubin < 1.5 x ULN (patients with Gilbert's disease exempt who should have bilirubin < 2x ULN)
    2. AST and ALT < 2.5 x upper limit of normal (ULN);
    3. Serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥60 mL/min
    4. Absolute neutrophil count (ANC) > 1500/mm³ without growth factor support
    5. Platelets > 75 000 cells/mm³
    6. Hemoglobin ≥9 g/dL (which may be obtained by transfusion or growth factor support)
    7. FT4 hormone levels within normal range
13. No prior treatment on a nivolumab and/or ipilimumab trial;
14. No prior treatment with an anti-CTLA-4 or anti-PD-1/-L1 targeted therapy
15. No gastrointestinal abnormalities including:

    1. Inability to take oral medication.
    2. Requirement for intravenous alimentation.
    3. Prior surgical procedures affecting absorption including gastric resection.
    4. Treatment for active peptic ulcer disease in the past 6 months.
    5. Malabsorption syndromes.
    6. Active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy;
16. No evidence of pre-existing uncontrolled hypertension as documented by baseline blood pressure reading. The baseline systolic blood pressure reading must be ≤140 mm Hg, and the baseline diastolic blood pressure readings must be ≤90 mm Hg. If baseline blood pressure reading exceeds the inclusion values a second blood pressure reading (taken at least 1 hour apart) must be documented in order to confirm the absence of uncontrolled hypertension. Patients whose hypertension is controlled by antihypertensive therapies are eligible;
17. No concurrent treatment:

    1. In another therapeutic clinical trial;
    2. No requirement for permanent therapeutic anticoagulation therapy.
18. Subjects with active, known, or suspected autoimmune disease are not eligible. Subjects with type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll.
19. Subjects requiring systemic treatment with either corticosteroids (> 8 mg daily methylprednisolone equivalent) or other immunosuppressive medications within 14 days of study enrollment. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
20. Adequate venous access to undergo a leukapheresis procedure.
21. No active uncontrolled seizure disorder.
22. No myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure or any unstable arrhythmia, cerebrovascular accident or transient ischemic attack, within the 12 months prior to study drug administration. No current or recent (within 1 month) use of a thrombolytic agent or a thrombo-embolic event;
23. No known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness;
24. No serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment;
25. No history of a malignancy (other than glioma) except those treated with curative intent for skin cancer (other than melanoma) or in situ breast or cervical cancer or those treated with curative intent for any other cancer with no evidence of disease for 5 years;
26. No other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study;
27. No dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol;
28. Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to treatment.; Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception measures during the period of therapy which should be continued for 12 weeks after the last dose of nivolumab. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate; No pregnancy or breastfeeding; a) No contra-indication for neurosurgical resection of the glioblastoma recurrence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2026-11-17 (Estimated); Study Completion 2026-11-17 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 30 weeks
  Estimate the survival of patients who are free from confirmed tumor.
Overall Survival (OS) | an average of 1 year
  Estimate the survival of patients who are alive.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larkin J, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Sep 24;373(13):1270-1. doi: 10.1056/NEJMc1509660. No abstract available. PMID 26398076
- [Background] Postow MA, Chesney J, Pavlick AC, Robert C, Grossmann K, McDermott D, Linette GP, Meyer N, Giguere JK, Agarwala SS, Shaheen M, Ernstoff MS, Minor D, Salama AK, Taylor M, Ott PA, Rollin LM, Horak C, Gagnier P, Wolchok JD, Hodi FS. Nivolumab and ipilimumab versus ipilimumab in untreated melanoma. N Engl J Med. 2015 May 21;372(21):2006-17. doi: 10.1056/NEJMoa1414428. Epub 2015 Apr 20. PMID 25891304
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Motzer RJ, Rini BI, McDermott DF, Redman BG, Kuzel TM, Harrison MR, Vaishampayan UN, Drabkin HA, George S, Logan TF, Margolin KA, Plimack ER, Lambert AM, Waxman IM, Hammers HJ. Nivolumab for Metastatic Renal Cell Carcinoma: Results of a Randomized Phase II Trial. J Clin Oncol. 2015 May 1;33(13):1430-7. doi: 10.1200/JCO.2014.59.0703. Epub 2014 Dec 1. PMID 25452452
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Topalian SL, Sznol M, McDermott DF, Kluger HM, Carvajal RD, Sharfman WH, Brahmer JR, Lawrence DP, Atkins MB, Powderly JD, Leming PD, Lipson EJ, Puzanov I, Smith DC, Taube JM, Wigginton JM, Kollia GD, Gupta A, Pardoll DM, Sosman JA, Hodi FS. Survival, durable tumor remission, and long-term safety in patients with advanced melanoma receiving nivolumab. J Clin Oncol. 2014 Apr 1;32(10):1020-30. doi: 10.1200/JCO.2013.53.0105. Epub 2014 Mar 3. PMID 24590637
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Eggermont AM, Chiarion-Sileni V, Grob JJ, Dummer R, Wolchok JD, Schmidt H, Hamid O, Robert C, Ascierto PA, Richards JM, Lebbe C, Ferraresi V, Smylie M, Weber JS, Maio M, Konto C, Hoos A, de Pril V, Gurunath RK, de Schaetzen G, Suciu S, Testori A. Adjuvant ipilimumab versus placebo after complete resection of high-risk stage III melanoma (EORTC 18071): a randomised, double-blind, phase 3 trial. Lancet Oncol. 2015 May;16(5):522-30. doi: 10.1016/S1470-2045(15)70122-1. Epub 2015 Mar 31. PMID 25840693
- [Background] Fransen MF, van der Sluis TC, Ossendorp F, Arens R, Melief CJ. Controlled local delivery of CTLA-4 blocking antibody induces CD8+ T-cell-dependent tumor eradication and decreases risk of toxic side effects. Clin Cancer Res. 2013 Oct 1;19(19):5381-9. doi: 10.1158/1078-0432.CCR-12-0781. Epub 2013 Jun 20. PMID 23788581
- [Background] Marabelle A, Kohrt H, Levy R. Intratumoral anti-CTLA-4 therapy: enhancing efficacy while avoiding toxicity. Clin Cancer Res. 2013 Oct 1;19(19):5261-3. doi: 10.1158/1078-0432.CCR-13-1923. Epub 2013 Aug 21. PMID 23965900
- [Background] Robert L, Harview C, Emerson R, Wang X, Mok S, Homet B, Comin-Anduix B, Koya RC, Robins H, Tumeh PC, Ribas A. Distinct immunological mechanisms of CTLA-4 and PD-1 blockade revealed by analyzing TCR usage in blood lymphocytes. Oncoimmunology. 2014 Jun 25;3:e29244. doi: 10.4161/onci.29244. eCollection 2014. PMID 25083336
- [Background] Preusser M, Lim M, Hafler DA, Reardon DA, Sampson JH. Prospects of immune checkpoint modulators in the treatment of glioblastoma. Nat Rev Neurol. 2015 Sep;11(9):504-14. doi: 10.1038/nrneurol.2015.139. Epub 2015 Aug 11. PMID 26260659
- [Background] Bouffet E, Larouche V, Campbell BB, Merico D, de Borja R, Aronson M, Durno C, Krueger J, Cabric V, Ramaswamy V, Zhukova N, Mason G, Farah R, Afzal S, Yalon M, Rechavi G, Magimairajan V, Walsh MF, Constantini S, Dvir R, Elhasid R, Reddy A, Osborn M, Sullivan M, Hansford J, Dodgshun A, Klauber-Demore N, Peterson L, Patel S, Lindhorst S, Atkinson J, Cohen Z, Laframboise R, Dirks P, Taylor M, Malkin D, Albrecht S, Dudley RW, Jabado N, Hawkins CE, Shlien A, Tabori U. Immune Checkpoint Inhibition for Hypermutant Glioblastoma Multiforme Resulting From Germline Biallelic Mismatch Repair Deficiency. J Clin Oncol. 2016 Jul 1;34(19):2206-11. doi: 10.1200/JCO.2016.66.6552. Epub 2016 Mar 21. PMID 27001570
- [Derived] Duerinck J, Lescrauwaet L, Dirven I, Del'haye J, Stevens L, Geeraerts X, Vaeyens F, Geens W, Brock S, Vanbinst AM, Everaert H, Caljon B, Bruneau M, Lebrun L, Salmon I, Kockx M, Tuyaerts S, Neyns B. Intracranial administration of anti-PD-1 and anti-CTLA-4 immune checkpoint-blocking monoclonal antibodies in patients with recurrent high-grade glioma. Neuro Oncol. 2024 Dec 5;26(12):2208-2221. doi: 10.1093/neuonc/noae177. PMID 39406392
- [Derived] Arrieta VA, Duerinck J, Burdett KB, Habashy KJ, Geens W, Gould A, Schwarze JK, Dmello C, Kim KS, Saganty R, Chen L, Moscona A, McCord M, Lee-Chang C, Horbinski CM, Zhang H, Stupp R, Neyns B, Sonabend AM. ERK1/2 Phosphorylation Predicts Survival in Recurrent Glioblastoma Following Intracerebral and Adjuvant PD-1/CTLA-4 Immunotherapy: A REMARK-guided Analysis. Clin Cancer Res. 2024 Jan 17;30(2):379-388. doi: 10.1158/1078-0432.CCR-23-1889. PMID 37939133
- [Derived] Duerinck J, Schwarze JK, Awada G, Tijtgat J, Vaeyens F, Bertels C, Geens W, Klein S, Seynaeve L, Cras L, D'Haene N, Michotte A, Caljon B, Salmon I, Bruneau M, Kockx M, Van Dooren S, Vanbinst AM, Everaert H, Forsyth R, Neyns B. Intracerebral administration of CTLA-4 and PD-1 immune checkpoint blocking monoclonal antibodies in patients with recurrent glioblastoma: a phase I clinical trial. J Immunother Cancer. 2021 Jun;9(6):e002296. doi: 10.1136/jitc-2020-002296. PMID 34168003